CLINICAL TRIAL: NCT00377546
Title: Comparison of Vitreous Levels of Acular LS 0.04%, Xibrom 0.09%, and Nevanac 0.1%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 5264
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Vitrectomy
Keywords: Retinal Surgery
MeSH Terms: interventions — nepafenac; bromfenac

INTERVENTIONS:
Drug: Nepafenac
Drug: Ketorolac LS, Bromfenac

SUMMARY:
To compare the penetration of three different NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Males or females scheduled to undergo Vitrectomy surgery
* Likely to complete all study visits and able to provide informed consent
* Visual potential of 20/25 or better

Exclusion Criteria:

* Known contraindications to any study medication or ingredients
* Active ocular diseases or uncontrolled systemic disease
* Active ocular allergies

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States